CLINICAL TRIAL: NCT06208592
Title: Comparative Study of Sedative Requirement Using Sevoflurane With Anaconda Device Versus Conventional Sedation in Patients With COVID-19
Brief Title: Comparative Study of Anaconda System Use Versus Conventional Sedation in COVID-19 Patients.
Status: Completed | Type: Observational
Sponsor: Hospital Español de Mexico (Other)
Collaborators: Universidad Nacional Autonoma de Mexico (Other)
Responsible Party: Principal Investigator, Jose J Zaragoza, MD, Dr., Hospital H+ Queretaro
Other Study IDs: 2020-01-Anaconda
Record Dates: First submitted 2024-01-15; First posted 2024-01-17 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: COVID-19; Respiratory Failure
Keywords: sedatives; acute kidney injury; SARS-CoV-2; mechanical ventilation
MeSH Terms: conditions — COVID-19; Respiratory Insufficiency; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Anaconda Group: Use of Anaconda devide at any point during the initial follow up (7 days) additional of conventional intravenous sedation
  Interventions: Device: Sevoflurane with AnaConDa
- Non-Anaconda Group: Use on conventional intravenous sedation, not using Anaconda device

INTERVENTIONS:
Device: Sevoflurane with AnaConDa — Sevoflurane administered with AnaConDa device
  Groups: Anaconda Group

SUMMARY:
At the beginning of 2020, a global alert emerged which saturated intensive care units due to COVID-19 worldwide. This caused a need for mechanical ventilation due to atypical pneumonias that had a rapid evolution and respiratory failure; therefore the consumption of sedative agents in the intensive care units escalated. Suboptimal sedation in the intensive care unit, increases the adverse effects, costs, and morbidity. For the time being, they focus on the use of intravenous agents such as propofol or dexmedetomidine, which are associated with tolerance, withdrawal, delirium, and hemodynamic effects. Consequently, the need arises to maximize availability and effectiveness, which is why the intervention of the ANACONDA conservation device is carried out, which works with a heat and humidity exchange filter capable of administering isoflurane or sevoflurane with an efficiency of 90%.

DETAILED DESCRIPTION:
Analyze the difference in intravenous sedation requirements in patients with COVID-19. Patients who were assisted by a mechanical ventilator with sevoflurane versus conventional sedation.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with confirmed COVI-19 infection and assited with mechanical ventilation who entered critical care department.

Exclusion Criteria:

* Tranfers to a different hospital.
* Death within the first 24 hours of hospital stay.

Ages: 27 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with confired COVID-19 infection assited with mechanical ventilation that required sedation.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2020-05-30 (Actual); Primary Completion 2020-09-18 (Actual); Study Completion 2020-11-06 (Actual)

PRIMARY OUTCOMES:
Intravenous sedation requirements | 7 days
  Amount of intravenous sedation required

SECONDARY OUTCOMES:
Delirium | Hospital stay (up to 30 days)
  Number of patients that suffered delirium
Acute kidney injury | Hospital stay (up to 30 days)
  Number of patients that suffered delirium
VAP | Hospital stay (up to 30 days)
  Number of patients that suffered ventilation acquired pneumonia

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Lomeli, MD, Study Chair — Hospital H+ Queretaro
Locations (1):
- Hospital H+ Queretaro, Querétaro City, Querétaro, Mexico

IPD SHARING:
Plan to Share IPD: Yes
Complete database will be shared as requested by the publishing journal, once the study is apporved.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Available one year after
Access Criteria: Journal provided